CLINICAL TRIAL: NCT07135284
Title: Real Life Evaluation of the LibAirty Airway Clearance System in Adults With Bronchiectasis (RELACS) - A Prospective Study
Brief Title: Real Life Evaluation of the LibAirty Airway Clearance System in Adults With Bronchiectasis (RELACS)
Status: Not yet recruiting | Type: Observational
Sponsor: Synchrony-Medical, Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: CL-00010
Record Dates: First submitted 2025-06-26; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Bronchiectasis Adult

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Adults with bronchiectasis: Adults with bronchiectasis, prescribed with the LibAirty airway clearance system
  Interventions: Device: Airway clearance system

INTERVENTIONS:
Device: Airway clearance system — The device is prescribed as part of each participant's regular medical care, independently of the study. The study does not assign the device or alter standard treatment. Participants are observed while using the device as part of their usual care.

SUMMARY:
The purpose of this study is to collect data to assess the use of the LibAirty™ System for improving bronchiectasis symptoms and healthcare resource utilization when it is used at home.

The main question this study is trying to answer is: How often do adults with bronchiectasis experience pulmonary exacerbations (flare-ups of their lung condition) while using the LibAirty™ airway clearance system at home?

Participants will use the LibAirty™ airway clearance system at home as prescribed by their doctor - the device is not being provided as part of the study. The study will last for 12 months from the time participants begin using LibAirty.

During the study period, participants will continue with their usual clinic visits. At some of these regular visits (up to 4 times over the year), participants will be asked to complete short questionnaires about their bronchiectasis symptoms and their experience using LibAirty. At these same visits, the study team will also review participants' medical records and collect information related to their bronchiectasis condition, such as test results, medications, and any hospital or emergency room visits.

DETAILED DESCRIPTION:
This prospective, single-arm, open-label study aims to evaluate the real-world use of the LibAirty™ Airway Clearance System for airway clearance in adult patients with bronchiectasis in a home setting. The primary objective is to assess the rate of pulmonary exacerbations during the 12-month study period, compared to the 12 months prior to enrollment, using each participant as their own historical control.

Importantly, this study is observational in nature. Participants are prescribed the LibAirty™ system by their treating physician as part of routine clinical care, independent of study enrollment. The study does not assign participants to receive the device, nor does it provide the device as part of the study. Participants will use the LibAirty™ system in the same manner and frequency as they would outside of the study, based on the physician's clinical judgment and standard treatment protocols.

The study will observe clinical outcomes in participants who are already prescribed the device. Data will be collected prospectively during regularly scheduled clinic visits that occur as part of each participant's standard care. At up to four of these visits, information will be gathered from medical records, and participants will complete validated questionnaires to assess health-related quality of life and user satisfaction with the LibAirty™ system. Adherence to therapy will be assessed using usage logs recorded by the device.

Additional clinical outcomes such as hospitalizations, emergency department visits, use of antibiotics for exacerbations, pulmonary function test results, and healthcare resource utilization related to bronchiectasis will be monitored. No investigational procedures, treatments, or interventions are introduced or modified by the study team.

This study is designed to generate real-world evidence on the effectiveness, adherence, and patient experience associated with the LibAirty™ system when used as part of standard bronchiectasis care in the home setting.

ELIGIBILITY:
Inclusion Criteria:

1. Have a radiological diagnosis of Bronchiectasis based on high resolution chest CT scan
2. Have bronchiectasis characterized by either:

   * Daily productive cough (as determined by a treating physician)
   * OR Available documentation from the last 12 months of 2 or more pulmonary exacerbations requiring antibiotic therapy
3. Be at age ≥ 21 years
4. Prescribed and receives the LibAirty system for home use
5. Be on a standard of care treatment plan that includes at least one physician encounter every 6 months
6. No change in treatment for Bronchiectasis in the 2-month period prior to enrollment
7. Signed informed consent

Exclusion Criteria:

1. Inability to independently perform therapy with the LibAirty system as directed
2. Any other condition that, in the opinion of the PI, could jeopardize the safety of the subject or impact the validity of the study results.
3. Pregnancy or planned pregnancy during the expected duration of the trial (12 months).

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with bronchiectasis who have been prescribed the LibAirty airway clearance system as part of their standard care. Participants will be identified and recruited from outpatient pulmonary or respiratory clinics affiliated with participating study sites.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-08-31 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint for this study is the rate of pulmonary exacerbations (PE). | 12 months

SECONDARY OUTCOMES:
Rate of respiratory related hospitalizations, including length of stay | 12 months
Rate of severe PEs (requiring IV antibiotics and/or hospitalization) | 12 months
Number of respiratory related ED visits | 12 months
Change from Baseline in PFTs (FEV1) | 12 months
Change from Baseline in PFTs (FVC) | 12 months
Change from Baseline in PFTs (FEV1/FVC) | 12 months
Change from baseline in Quality of Life (QoL-B) | 12 months
User satisfaction with the LibAirty system | 12 months
  Evaluated using a LibAirty™ system user satisfaction questionnaire
Adherence to therapy | 12 months
  Adherence to therapy will be evaluated using device usage logs
Healthcare resource utilization resulting from respiratory condition | 12 months
  Cost of treatments, hospitalizations and ED visits

OTHER OUTCOMES:
Time to first PE and median time between PEs | 12 months
Percent of patients who have not experienced a PE for 6 months and 12 months | 6 months and 12 months
Number of courses of antibiotics prescribed for pulmonary exacerbations, including duration and route of administration | 12 months